CLINICAL TRIAL: NCT01310192
Title: Cancer Localization in the Prostate With F-18 Fluorocholine Positron Emission Tomography
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Queen's Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RA-2004-040; PC04130
Record Dates: First submitted 2009-06-24; First posted 2011-03-08 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Investigational Imaging Device
  Interventions: Device: Fluourine-18 Fluoromethylcholine PET/CT Imaging

INTERVENTIONS:
Device: Fluourine-18 Fluoromethylcholine PET/CT Imaging — Single-dose Study
  Other Names: 18F-choline PET/CT; Fluorocholine PET/CT

SUMMARY:
The purpose of this project is to develop and evaluate fluorine-18 (F-18) fluorocholine (FCH) positron emission tomography (PET) as an imaging technique that can be used to delineate malignant tumors in the prostate gland. The proposed technique works by measuring the tissue metabolism of FCH, a substrate that is preferentially metabolized by cancer cells due to malignant over-expression of the choline transporter and choline kinase enzyme. The project scope covers a clinical study to recruit men with prostate cancer who have elected treatment by radical prostatectomy surgery. These men will undergo pre-operative PET scanning to measure F-18 FCH uptake in anatomical sextants of the prostate gland. Imaging results will be compared to histopathologic analyses of the prostatectomy specimen to determine the accuracy of F-18 FCH PET for detecting cancerous prostate sextants.

ELIGIBILITY:
Inclusion Criteria:

* Clinically Organ Confined Prostate Cancer Electing Radical Prostatectomy

Exclusion Criteria:

* Weight > 300 lb

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Histopathologic Diagnosis - sextant diagnosis by whole-prostate step section histopathologic analysis | Immediate - no longitudinal data collected

CONTACTS AND LOCATIONS:
Locations (1):
- Tripler Army Medical Center, Tripler AMC, Hawaii, United States

REFERENCES:
- [Background] DeGrado TR, Kwee SA, Coel MN, Coleman RE. The impact of urinary excretion of (18)F-labeled choline analogs. J Nucl Med. 2007 Jul;48(7):1225. doi: 10.2967/jnumed.107.040667. No abstract available. PMID 17607041
- [Background] Kwee SA, Coel MN, Lim J, Ko JP. Prostate cancer localization with 18fluorine fluorocholine positron emission tomography. J Urol. 2005 Jan;173(1):252-5. doi: 10.1097/01.ju.0000142099.80156.85. PMID 15592091
- [Result] Kwee SA, Thibault GP, Stack RS, Coel MN, Furusato B, Sesterhenn IA. Use of step-section histopathology to evaluate 18F-fluorocholine PET sextant localization of prostate cancer. Mol Imaging. 2008 Jan-Feb;7(1):12-20. PMID 18384719
- [Result] Kwee SA, DeGrado TR, Talbot JN, Gutman F, Coel MN. Cancer imaging with fluorine-18-labeled choline derivatives. Semin Nucl Med. 2007 Nov;37(6):420-8. doi: 10.1053/j.semnuclmed.2007.07.003. PMID 17920349